CLINICAL TRIAL: NCT01347684
Title: Assessing the Effectiveness of Two Treatment Strategies for Tension-type Headache
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI left University of Minnesota
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1103M96812
Record Dates: First submitted 2011-04-28; First posted 2011-05-04 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Tension-type Headache
Keywords: headache; elavil; splints; physical therapy; behavioral therapy
MeSH Terms: conditions — Tension-Type Headache; Headache | interventions — Behavior Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care using current drugs (Active Comparator): Standard care with drug intervention
  Interventions: Drug: Standard care using current drugs
- Behavioral therapy, splint therapy and physical therapy (Experimental): Using rehabilitation for comparing use of drug
  Interventions: Behavioral: Behavioral therapy, splint therapy and physical therapy

INTERVENTIONS:
Behavioral: Behavioral therapy, splint therapy and physical therapy — Includes patient education, use of a mouth guard, jaw muscle exercises and brief cognitive-behavioral intervention.
  Other Names: Medications: Amitryptoline or has unacceptable side-effects, then other tricyclics and/or muscle relaxants are allowed.1
  Arms: Behavioral therapy, splint therapy and physical therapy
Drug: Standard care using current drugs — Standard Drug therapy
  Arms: Standard care using current drugs

SUMMARY:
The primary aim of the pilot data proposal is to compare usual care (medications) versus multi-disciplinary treatment in temporomandibular disorder (TMD) patients.

DETAILED DESCRIPTION:
The primary aim of the pilot data proposal is to compare usual care (medications) versus multi-disciplinary treatment in TMD patients with episodic or chronic tension-type headache (TTH) with pericranial tenderness involving the temporalis muscle at reducing the intensity of TTH pain at 1 and 6 months. The hypothesis is that a team approach will reduce the intensity of headache more than usual care in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

Fifty consecutive subjects (Age 18 to 65) will be included when they fulfill the diagnostic criteria for episodic or chronic TTH with pericranial muscle tenderness3 and TMD including myofascial pain involving the temporalis muscle -

Exclusion Criteria:

Exclusion criteria, assessed by review of medical history, include:

* systemic rheumatic disease
* widespread pain
* pregnancy
* concurrent use of tricyclic antidepressants, steroids, anti-inflammatories, muscle relaxants, or narcotics
* major psychiatric disease
* any medical contraindications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline of headache intensity of pain using pain scale of 1-10 | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Schiffman, DDS, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota School of Dentistry, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota